CLINICAL TRIAL: NCT06766331
Title: Integrating Infectious Diseases Screening and Treatment With Medication Assisted Therapy for Veterans With Opioid Use Disorder
Brief Title: Integrated Care Versus Usual Care for Opioid Use Disorder and Infectious Diseases in Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: INFA-010-24S; 1IK2CX002822-01A1 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; HIV; Hepatitis C Virus; Gonorrhea; Chlamydia; Syphilis; Sexually Transmitted Infection; Integrated Care; Medications for Opioid Use Disorder
Keywords: Hepatitis C; HIV; sexually transmitted diseases; Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Hepatitis C; Gonorrhea; Chlamydia Infections; Syphilis; Sexually Transmitted Diseases | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either integrated care (infectious diseases screening and/or PrEP for HIV plus opioid use disorder clinical care within one clinic appointment) or treatment as usual (opioid use disorder clinical care plus infectious diseases clinic referral for testing and/or PrEP for HIV)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated care (Experimental): Study visit 1: Participants will first complete a study interview, then will receive a prescription for laboratory testing for HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), gonorrhea, chlamydia, and syphilis. Those who meet eligibility criteria for PrEP will receive a prescription for PrEP (emtricitabine 200 mg (FTC)/25 mg tenofovir alafenamide-emtricitabine (TAF) or once daily emtricitabine 200 mg (FTC)/300 mg tenofovir disoproxil fumarate-emtricitabine (TDF)), and will be referred to the Infectious Diseases clinic for PrEP follow-up. Participants will then complete a standard SUD clinic appointment. Study visit 2: Participants will follow-up at 90 days in the SUD clinic where they will repeat the study interview, followed by receipt of standard SUD clinical care.
  Interventions: Other: Integrated care
- Treatment as usual (No Intervention): Study visit 1: Participants will first complete a study interview, then will complete a standard SUD clinic appointment. After the SUD appointment, participants will be referred to the Infectious Diseases clinic to receive standard infectious diseases laboratory testing, including HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), gonorrhea, chlamydia, and syphilis. Those who meet eligibility criteria for PrEP will receive a prescription for PrEP (emtricitabine 200 mg (FTC)/25 mg tenofovir alafenamide-emtricitabine (TAF) or once daily emtricitabine 200 mg (FTC)/300 mg tenofovir disoproxil fumarate-emtricitabine (TDF) through the infectious diseases clinic. Study visit 2: Participants will follow-up at 90 days in the SUD clinic where they will repeat the study interview, followed by receipt of their standard SUD clinical care.

INTERVENTIONS:
Other: Integrated care — Receipt of infectious diseases laboratory testing and/or PrEP for HIV within a single substance use disorder clinic appointment.
  Arms: Integrated care

SUMMARY:
Opioid use disorder (OUD) confers a higher risk of acquiring and transmitting infectious diseases, which may have long-term health consequences in Veterans. Treatment of OUD with medication assisted therapy is highly effective, however this often occurs independently of infectious diseases care. This project will test out a new model that combines infectious diseases and OUD care within one VA clinic appointment. This new care model may improve the health of Veterans and reduce cost and time required for Veterans who often need to attend multiple outpatient appointments.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) is associated with increased risk for overdose as well as acquisition and transmission of infectious diseases (ID), including HIV, hepatitis C virus (HCV), and bacterial sexually transmitted infections (STI). Previous studies support improved clinical outcomes when integrating treatment for OUD and screening and treatment of HIV and HCV in non-Veteran populations. However, clinical care for Veterans with OUD often requires appointments with multiple different healthcare providers. These care silos place an increased burden on this patient population who often have barriers to appointment attendance. Improved integration OUD and ID clinical care is needed. In a recent study of Veterans with OUD who accessed care at the Northport VA (Long Island, NY) the investigators identified 216 (43%) Veterans who had a history of injecting drug use and of those, 134 (62%) had HCV and 30 (13.9%) had at least one severe injection related infection requiring hospitalization. The investigators also found low rates of screening for bacterial sexually transmitted infections, including syphilis (n=371, 74%), gonorrhea (n=160, 31.9%), chlamydia (n=169, 33.7%) and low uptake of HIV pre-exposure prophylaxis (PrEP) (n=4, 0.8%). In this pilot study, the investigators will assess the feasibility and acceptability of an integrated ID screening and PrEP intervention for Veterans with OUD who are engaged in care through the Northport VA SUD clinic. The investigators will randomize Veterans to receive either integrated care (HIV, HCV, STI screening and/or PrEP plus SUD care) or treatment as usual (SUD care plus ID clinic referral). The investigators will also compare rates of HIV, HCV and bacterial STI screening as well as PrEP uptake between the groups. This research will benefit male and female Veterans with OUD. This project will be carried out at the Northport Veterans Affairs Medical Center (NVAMC). Information obtained from this study will be utilized to inform a larger multi-site VA trial assessing the efficacy of IC versus usual care.

ELIGIBILITY:
Inclusion Criteria:

* US Veteran
* Able to provide written informed consent in English
* Living in the community (Nassau, Suffolk, Kings, Queens, Bronx, Westchester, Rockland counties, NY)
* Documented diagnosis of moderate to severe opioid use disorder
* Seeking care at the Northport VA substance use disorder clinic for opioid use disorder treatment
* Willing to have HIV, HBV, HCV, or bacterial STI testing to determine negative or positive status
* Persons who test negative for HIV need to meet CDC PrEP eligibility criteria in the 6 months prior to enrollment

Exclusion Criteria:

* Severe medical or psychiatric disability making participation unsafe
* Unable to provide written consent
* PrEP exclusion: HIV positive test; HBV positive test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2028-04-03 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Infectious diseases screening uptake during intervention period | 90 days
  Proportion of Veterans who completed any screening for HIV, hepatitis C virus (HCV), gonorrhea, chlamydia, or syphilis during the intervention period

SECONDARY OUTCOMES:
PrEP uptake during intervention period | 90 days
  Proportion who initiated PrEP for HIV during the intervention period
HIV screening uptake during intervention period | 90 days
  Proportion who completed screening for HIV during the intervention period
HCV screening uptake during intervention period | 90 days
  Proportion who completed screening for HCV during the intervention period
Gonorrhea screening uptake during intervention period | 90 days
  Proportion who completed screening for gonorrhea during the intervention period
Chlamydia screening uptake during intervention period | 90 days
  Proportion who completed screening for chlamydia during the intervention period
Syphilis screening uptake during intervention period | 90 days
  Proportion who completed screening for syphilis during the intervention period
PrEP uptake during follow-up period | 270 days
  Proportion who initiated PrEP for HIV at any point during the follow-up period
HIV screening uptake during follow-up period | 270 days
  Proportion who completed screening for HIV at any point during the follow-up period
HCV screening uptake during follow-up period | 270 days
  Proportion who completed screening for HCV at any point during the follow-up period
Gonorrhea screening uptake during follow-up period | 270 days
  Proportion who completed screening for gonorrhea at any point during the follow-up period
Chlamydia screening uptake during follow-up period | 270 days
  Proportion who completed screening for chlamydia at any point during the follow-up period
Syphilis screening uptake during follow-up period | 270 days
  Proportion who completed screening for syphilis at any point during the follow-up period
PrEP retention during the intervention period | 90 days
  Proportion of Veterans who adhered to the PrEP prescription during the intervention period
PrEP retention during the follow-up period | 270 days
  Proportion of Veterans who adhered to the PrEP prescription during the follow-up period

OTHER OUTCOMES:
Feasibility of the integrated care intervention | 90 days
  Proportion of Veterans who agreed that the integrated care intervention was a feasible care model for the substance use disorder clinic
Acceptability of the integrated care intervention | 90 days
  Proportion of Veterans who agreed that the integrated care intervention was an acceptable care model for the substance use disorder clinic

CONTACTS AND LOCATIONS:
Overall Officials: Audun J Lier, MD, Principal Investigator — Northport VA Medical Center, Northport, NY
Locations (1):
- Northport VA Medical Center, Northport, NY, Northport, New York, United States

IPD SHARING:
Plan to Share IPD: No